CLINICAL TRIAL: NCT01820910
Title: International Prospective Phase 2 Trial Addressing the Efficacy of First-line Chlamydophila Psittaci-eradicating Therapy With Protracted Administration of Doxycycline Followed by Eradication Monitoring and Antibiotic Re-treatment at Infection Re-occurrence in Patients With Newly Diagnosed Ocular Adnexal Marginal Zone Lymphoma (OAMZL)
Brief Title: Phase II Trial of First-line Doxycycline for Ocular Adnexal Marginal Zone Lymphoma Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG39
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Marginal Zone Lymphoma of Ocular Adnexal
MeSH Terms: interventions — Doxycycline

ARMS (1):
- Doxycycline (Experimental)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — All enrolled patients will be treated with doxycycline 100 mg bid daily, orally, for four weeks followed by four weeks rest, repeated for three cycles. Response will be assessed by MRI (magnetic resonance imaging) and ophthalmologic examination at the end of the planned treatment. Patients who will achieve complete response, partial response or have a stable disease at 3 months from upfront doxycycline will be monitored for infection re-occurrence and assessed for response with MRI and ophthalmologist evaluation every six months for the first five years.

SUMMARY:
Objective of this trial is to establish the efficacy of an upfront targeted therapy consisting of Chlamydophila psittaci (Cp)-eradicating therapy with prolonged administration of doxycycline followed by eradication monitoring and antibiotic re-treatment at infection re-occurrence in patients with newly diagnosed ocular adnexae marginal zone lymphoma The primary endpoint is the 2-year progression-free survival (PFS) of patients with newly diagnosed stage-IE lymphoma treated with the experimental strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of marginal zone lymphoma of the ocular adnexae (OAMZL)
2. Single or bilateral lesion (stage IE) localised to the ocular adnexae (conjunctiva, lachrymal gland or sac, orbit soft tissue, eyelid)
3. Absence of B symptoms
4. Previously untreated patients
5. No systemic antibiotic therapy in the last three months before enrolment
6. Age >18 years
7. ECOG PS 0-2
8. Negative HIV, HBV and HCV serology
9. Adequate bone marrow, renal, and hepatic function
10. No previous or concurrent malignancies with the exception of surgically cured carcinoma in situ of the cervix, carcinoma of the skin or other cancers without evidence of disease at least from 5 years
11. Absence of any familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
12. Sexually active patients of childbearing potential must implement adequate contraceptive measures during study participation
13. No concurrent treatment with other experimental drugs
14. Patient-signed informed consent obtained before registration

Exclusion Criteria:

1. Pregnant or lactating women
2. Known allergy to tetracycline
3. Patients unwilling to comply with the requirements of follow-up
4. Myasthenia gravis (tetracycline can exacerbate muscle weakness)
5. Systemic lupus erythematous (tetracycline can exacerbate this condition)
6. Patients with large or rapidly enlarging tumors requiring immediate radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 2-year from start of treatment
  from the date of the start of treatment to relapse, progression or death, or to the last date of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Ferreri, MD, Study Chair — Ospedale San Raffaele, Milan, Italy
Locations (7):
- Italy (7):
  - AO Ospedali Riuniti Papardo Piemonte, Messina
  - Ospedale San Raffaele, Milan
  - Ematologia, Parma
  - Ospedale Civile, Piacenza
  - Università La Sapienza, Rome
  - Molinette 1, Torino
  - Ospedale dell'Angelo, Venezia